CLINICAL TRIAL: NCT05208996
Title: An Open-safety Study of the siCoV/KK46 Drug Administered Via an Inhaled Route in Healthy Volunteers
Brief Title: The siCoV/KK46 Drug Open-safety Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Research Center - Institute of Immunology Federal Medical-Biological Agency of Russia (Other)
Collaborators: St. Petersburg Research Institute of Vaccines and Sera (Other Government)
Responsible Party: Principal Investigator, Latysheva Tatyana, The Head of Immunopathology Department, National Research Center - Institute of Immunology Federal Medical-Biological Agency of Russia
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SiCoV/KK46-2020
Record Dates: First submitted 2021-11-30; First posted 2022-01-26 (Actual); Last update posted 2022-01-26 (Actual); Status verified 2022-01

CONDITIONS: COVID-19
Keywords: COVID-19; siRNA; SARS-CoV-2
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: This is a dose-escalation trial, all participants will receive single or multiple treatment with siCoV/KK46 via an inhaled route. Participants enrolled in this trial may receive one of the following doses:
  Cohort 1: 3.7 mg; Cohort 2: 11.1 mg; Cohort 3: 22.2 mg
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- siCoV/KK46 (Experimental): Drug contains anti-SARS-CoV-2 siRNAs/KK-46 (peptide dendrimer) complexes for inhalation use
  Interventions: Drug: siCoV/KK46

INTERVENTIONS:
Drug: siCoV/KK46 — The modified phase I "3 + 1+1" study design was used in dose escalation from low dose to high dose to determine the maximum daily dose. Sequential assignment of Patient cohorts to one of three dose levels of inhaled siCoV/KK46: 3.7 mg, 11.1 mg, 22.2 mg.

SUMMARY:
This is an open-label, dose-escalation phase I study to assess the safety and tolerability of siCoV/KK46 in healthy volunteers. The purpose of this study is to determine the maximum daily dose of siCoV/KK46 as a single agent in adult healthy participants. Based on preclinical data from this institution, the investigators hypothesize that SARS-CoV-2 inhibition with siCoV/KK46 could potentially reduce pulmonary inflammation, thereby improving COVID-19 patient outcomes.

DETAILED DESCRIPTION:
This is an open-label, dose-escalation phase I study to assess the safety and tolerability of single and multiple doses of siCoV/KK46 in healthy male volunteers.

This study include 3 cohorts received 3.7 mg, 11.1 mg, 22.2 mg of the siCoV/KK46, respectively, via inhalation route.

All subjects will undergo scheduled safety and tolerability assessments while in the clinical unit and as outpatients to the end of the follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy men aged 18 to 45 years
2. Able to give informed consent and attend all study visits
3. Blood pressure level: systolic blood pressure 100 to 139 mm Hg, diastolic blood pressure 60 to 89 mm Hg.
4. Heart rate from 60 to 90 beats per minute
5. Body mass index 18.5 -30. The body weight should be ≥ 55 kg;
6. Men must agree to use the reliable contraception while on study medication and for posttrial contraception for 30 days
7. Be able to understand and comply with protocol requirements

Exclusion Criteria:

1. A burdened allergic history.
2. Previous adverse reactions to the active substance and/or excipients included in the drug.
3. Chronic diseases of the cardiovascular, lymphatic, respiratory, nervous, endocrine, digestive, musculoskeletal, integumentary, immune systems, as well as the genitourinary apparatus and hematopoietic organs.
4. Weakness of the inspiratory muscles of respiration (according to spirometry result).
5. Acute infectious diseases symptoms in the last 4 weeks before screening.
6. Treatment with any medicine that have a pronounced effect on hemodynamics and affects the liver function (barbiturates, omeprazole, cimetidine, etc.) within 2 months prior to screening.
7. Regular treatment with any medicine less than 2 weeks prior to screening and single treatment less than 7 days prior screening.
8. Donation of blood or plasma less than 3 months prior to screening.
9. Transfusion of blood and/or its components less than 3 months prior to screening.
10. Participation in other investigational drug or device clinical trials within 90 days prior to screening.
11. Drinking of more than 10 units of alcohol (1 unit of alcohol is equivalent to 330 mL of beer, 150 mL of wine or 40 mL of strong alcoholic drinks) per week within the last month prior to inclusion in the study and/or history of alcohol, drug or chemical abuse.
12. Smoking more than 10 cigarettes currently, or history of smoking this number of cigarettes within 6 months prior to screening.
13. Positive blood tests for HIV, hepatitis B and С, syphilis. Positive PCR test results for SARS-CoV-2(nasal swab).
14. Positive result on a urine drug screening test.
15. Positive test for ethanol vapor in exhaled air.
16. Planned hospitalization during the period of participation in the study, for any reason other than hospitalization specified by this protocol.
17. Inability or inability to follow the protocol, to perform the procedures prescribed by the protocol, to follow a diet, activity regime.
18. Any conditions that, according to the researcher's, may be a contraindication to the participation in the study.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2021-01-22 (Actual); Primary Completion 2021-03-26 (Actual); Study Completion 2021-03-26 (Actual)

PRIMARY OUTCOMES:
This is an open-label, dose-escalation phase I study to assess the safety and tolerability of siCoV/KK46 in healthy volunteers | Within 72 hours after single treatment with siCoV/KK46
  Adverse Events
Vital Signs | Within 72 hours after single treatment with siCoV/KK46
  Blood pressure in mm Hg
Body Temperature control | Within 72 hours after single treatment with siCoV/KK46
  Taking an Axillary Temperature
Heart rate | Within 72 hours after single treatment with siCoV/KK46
  Heart Rate in beats per minute
Clinical Chemistry to asses Potassium level | Within 72 hours after single treatment with siCoV/KK46
  Measurement of Potassium level in blood
Clinical Chemistry to asses Sodium level | Within 72 hours after single treatment with siCoV/KK46
  Measurement of Sodium level in blood
Clinical Chemistry to asses Chloride level | Within 72 hours after single treatment with siCoV/KK46
  Measurement of Chloride level in blood
Clinical Chemistry to asses Bicarbonate level | Within 72 hours after single treatment with siCoV/KK46
  Measurement of Bicarbonate level in blood
Clinical Chemistry to asses Calcium level | Within 72 hours after single treatment with siCoV/KK46
  Measurement of Calcium level in blood
Clinical Chemistry to asses Phosphate level | Within 72 hours after single treatment with siCoV/KK46
  Measurement of Phosphate level in blood
Clinical Chemistry to asses Creatine phosphokinase level | Within 72 hours after single treatment with siCoV/KK46
  Measurement of Creatine phosphokinase level in blood
Clinical Chemistry to asses Blood urea nitrogen level | Within 72 hours after single treatment with siCoV/KK46
  Measurement of Blood urea nitrogen level
Clinical Chemistry to asses Albumin level | Within 72 hours after single treatment with siCoV/KK46
  Measurement of Albumin level in blood
Clinical Chemistry to asses Protein level | Within 72 hours after single treatment with siCoV/KK46
  Measurement of Protein level in blood
Clinical Chemistry to asses Aspartate transaminase level | Within 72 hours after single treatment with siCoV/KK46
  Measurement of Aspartate transaminase level in blood
Clinical Chemistry to asses Alanine transaminase level | Within 72 hours after single treatment with siCoV/KK46
  Measurement of Alanine transaminase level in blood
Clinical Chemistry to asses Alkaline phosphatase level | Within 72 hours after single treatment with siCoV/KK46
  Measurement of Alkaline phosphatase level in blood
Clinical Chemistry to asses Bilirubin level | Within 72 hours after single treatment with siCoV/KK46
  Measurement of Bilirubin level in blood
Blood Glucose Test | Within 72 hours after single treatment with siCoV/KK46
  Measurement of Glucose level
Haematology blood test | Within 72 hours after single treatment with siCoV/KK46
  Qualitative and quantitative composition of the cellular components of the blood
Urinalysis | Within 72 hours after single treatment with siCoV/KK46
  Physical, chemical, and microscopic examination of urine
12-Lead Electrocardiogram | Within 72 hours after single treatment with siCoV/KK46
  Measurement of Heart rate; PR, QRS, RR, QT and QTc intervals from digital recordings

CONTACTS AND LOCATIONS:
Locations (1):
- NRC Institute of Immunology FMBA, Moscow, Russia